CLINICAL TRIAL: NCT02043743
Title: Autologous Stem Cells Transplantation in Patients With Idiopathic and Drug Induced Premature Ovarian Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: El-Rayadh Fertility Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT0221012014; RFC0221012014 (Other Grant/Funding Number: RFC0221012014)
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laboratory and Clinical (Experimental): Biological: Stem Cells 60 ml of bone marrow will aspirated and used for stem cells isolation. Then stem cells will cultured using autologous serum, characterized and prepared using GMP rules and finally injected into rete testis.
  Stem Cell Dose:
  •3-5 Million Autologous MSCs Injected into Ovarian tissue.
  Interventions: Biological: Biological: Stem Cells

INTERVENTIONS:
Biological: Biological: Stem Cells — Biological: Stem Cells 60 ml of bone marrow will aspirated and used for stem cells isolation. Then stem cells will cultured using autologous serum, characterized and prepared using GMP rules and finally 3-5 million MSCs injected into ovarian tissue.
  Other Names: Stem Cells Transplantation

SUMMARY:
Premature ovarian failure (POF), also known as premature ovarian insufficiency, primary ovarian insufficiency (this is the most accurate term as some women may still conceive), premature menopause, hypergonadotropic hypogonadism is defined as failure of the ovary to function adequately in a woman younger than 40 years, in its role either as an endocrine organ or as a reproductive organ, a condition characterized by amenorrhea, hypoestrogenism, and elevated serum gonadotropin levels (which demonstrate that the ovaries are no longer responding to circulating FSH by producing estrogen and developing fertile eggs) in women younger than 40 years. This condition occurs in approximately 1% of women and it has important physical and psychological consequences/impact in those patients.

The purpose of this study is to investigate the role of the transplantation of bone marrow derived stem cells into ovarian tissue for treatment of premature ovarian failure and to assess their ability to differentiate into germ cells.

DETAILED DESCRIPTION:
This study is an open-label investigation of the efficacy of injection of autologous adult bone marrow derived stem cells into the ovarian stroma of patients with premature ovarian failure. Sixty women with premature ovarian failure will be recruited in this study after a written informed consent. Diagnosis will be based mainly on history taking, physical examination and investigations. Laboratory investigations will include Serum follicle-stimulating hormone (FSH), serum estrogen measurement and serum AMH. The anterior pituitary secretes FSH and LH at high levels due to the dysfunction of the ovaries and consequent low estrogen levels. Typical FSH in POF patients is over 40 mlU/ml (post-menopausal range). Subjects will be enrolled based on specific inclusion/exclusion criteria and evaluated at regular post transplant intervals. Human adult bone marrow derived stem cells will be transplanted by a gynecological surgeon through a standard surgical approach (transvaginal U/S guided approach). Subjects will be monitored frequently for a total of one year after adult bone marrow stem cells cell injection. For safety of participants, Bone Marrow Stem cells will be injected in one ovary only and the other ovary will be spared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal karyotype spontaneous premature ovarian failure.
* Patients between 18 - 40 years old.

Exclusion Criteria:

* Patients with secondary ovarian failure (e.g. hypothalamic causes).
* Pregnancy and lactation.
* Autoimmune diseases.
* Those with major medical problems such as malignancy, hepatitis, etc.
* Abnormal karyotyping (e.g. turner syndrome, fragile X syndrome….).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Cases Improvement | 48 Weeks
  Decline in serum FSH level. Rise in serum estrogen level Elevation in serum AMH level

SECONDARY OUTCOMES:
Cases Improvement | 48 Weeks
  Disappearance of menopausal symptoms e.g. hot flashes Rise in serum AMH level. Pregnancy rate within 1 year. Miscarriage rate within one year of injection. Long term follow-up for any adverse effect, assessed for one year from injection.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. Hesham Elshaer, MD, Principal Investigator — El-Rayadh Fertility Center; Sayed Bakry, PhD, Study Director — Al-Azhar University; Wael Abu El Khier, MD, Study Chair — Military Academy; Hala Gabr, MD, Study Chair — Cairo University
Locations (1):
- El-Rayadh Fertility Center, Giza, Egypt